CLINICAL TRIAL: NCT02587793
Title: Kaohsiung Medical University Chung-Ho Memorial Hospital
Brief Title: Primary Culture of Residual Specimens Obtained From Aspiration of Hepatic Tumor to Predict the Prognosis of the Patients
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Zu-Yau Lin, Professor, Kaohsiung Medical University Chung-Ho Memorial Hospital
Other Study IDs: KMUH-IRB-20140182
Record Dates: First submitted 2015-10-24; First posted 2015-10-27 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; primary culture; fine-needle aspiration; cancer-associated fibroblast
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — If the cultured cells can become cell lines, these cell lines will be stored.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Barcelona Clinic Liver Cancer (BCLC) staging: The tumor stages of the patient are classified as BCLC stage 0, A, B, C, or D.
  Interventions: Other: not interventional study

INTERVENTIONS:
Other: not interventional study

SUMMARY:
The aim of this project is to investigate whether the proliferative speeds of cultured cells using our method can be integrated into Barcelona Clinic Liver Cancer (BCLC) staging classification for the possibility of personalized treatment and prediction the outcomes in hepatocellular carcinoma (HCC) patients.

DETAILED DESCRIPTION:
A total of at least 150 patients will be included and followed for at least one year. The proliferative speeds of cultured cells will be classified into (a) rapid proliferation of HCC cells with or without concomitant rapid proliferation of cancer-associated fibroblasts (CAFs), (b) rapid proliferation of CAFs alone, and (c) slow proliferation three groups. The definition for the rapid proliferation of cultured cells fits at least one of the following two items: (1) growth area of cultured cells at the 15th-28th day > two times of the growth area measured at the 14th day, or (2) growth area of cultured cells at the 15th-28th day > 70% growth area of the 25 cm flask. The GraphPad Prism software version 4.03 (GraphPad Software, Inc., La Jolla, CA, USA) is applied for statistical analysis. Influence of the proliferative speeds of cultured cells on survival and cancer progression will be calculated by the logrank test. The statistical significance is defined as P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are proven to have HCC based on fine-needle aspiration of the tumor.
2. Patient have residual specimens obtained from fine-needle aspiration of the tumor.
3. Patients agree to participate this study after fully explanation.

Exclusion Criteria:

1. Patients are not proven to have HCC based on fine-needle aspiration of the tumor.
2. Patient do not have residual specimens obtained from fine-needle aspiration of the tumor.
3. Patients do not agree to participate this study after fully explanation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are proven to have HCC based on fine-needle aspiration of the tumor and also have residual specimens for culture are included.
Sampling Method: Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2014-10; Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
survival | one year
  Correlation between the proliferative speeds of cultured cells and one year survival of the patients after aspiration of the tumor will be investigated.

SECONDARY OUTCOMES:
cancer progression | one year
  Correlation between the proliferative speeds of cultured cells and HCC progression one year after aspiration of the tumor will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Zu-Yau Lin, MD, Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (2):
- Taiwan (2):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital, Kaohsiung City

REFERENCES:
- [Result] Lin ZY, Chuang WL, Chuang YH, Yu ML, Hsieh MY, Wang LY, Tsai JF. Discordant influence of amphotericin B on epirubicin cytotoxicity in primary hepatic malignant cells collected by a new primary culture technique. J Gastroenterol Hepatol. 2006 Feb;21(2):398-405. doi: 10.1111/j.1440-1746.2005.04026.x. PMID 16509865
- [Result] Lin ZY, Wu CC, Chuang YH, Chuang WL. Clinical utility of a simple primary culture method in hepatocellular carcinoma patients. J Gastroenterol Hepatol. 2015 Feb;30(2):352-7. doi: 10.1111/jgh.12693. PMID 25087586